CLINICAL TRIAL: NCT04612010
Title: WAVES: Wobble-oscillator Auditory/Visual Excitatory Stimulation for Mal de Debarquement Syndrome
Brief Title: WAVES for Mal de Debarquement Syndrome
Acronym: WAVESMdDS
Status: Withdrawn | Phase: Early Phase 1 | Type: Interventional
Why Stopped: Hypothesis change
Sponsor: University of Minnesota (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Single | Purpose: Device Feasibility
Other Study IDs: NEUR-2020-29419
Record Dates: First submitted 2020-10-26; First posted 2020-11-02 (Actual); Last update posted 2023-05-09 (Actual); Status verified 2023-05

CONDITIONS: Mal de Debarquement Syndrome
MeSH Terms: conditions — Mal de debarquement

STUDY DESIGN:
Intervention Model Description: The participants will be in an n-of-1 design with each participant receiving each frequency of stimulation in a randomized blinded order.
Who Masked: Participant
Masking Description: Each arm involves real stimulation but only one is consistent with the hypothesis of desynchronization. The participant will not be aware of which administration is providing the target frequency of stimulation.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Alpha frequency (Active Comparator): Wobble oscillation will revolve the individual alpha frequency
  Interventions: Device: WAVES (Wobble-oscillator Auditory/Visual Excitatory Stimulation)
- Alpha frequency plus (Active Comparator): Wobble oscillation will revolve the individual alpha frequency plus 0.5Hz
  Interventions: Device: WAVES (Wobble-oscillator Auditory/Visual Excitatory Stimulation)
- Theta frequency (Sham Comparator): Wobble oscillation will revolve the individual theta frequency
  Interventions: Device: WAVES (Wobble-oscillator Auditory/Visual Excitatory Stimulation)

INTERVENTIONS:
Device: WAVES (Wobble-oscillator Auditory/Visual Excitatory Stimulation) — An app-based stimulation program administered that provides desynchronizing visual and auditory stimulation. The frequency of the stimulation oscillates around the baseline frequency determined by EEG.
  Other Names: WAVES

SUMMARY:
This study will be recruiting individuals with Mal de Debarquement Syndrome (MdDS), a disorder caused by entrainment to oscillating motion that leads to persistent oscillating vertigo. The typical triggers for MdDS are sea and air travel. Prior studies on MdDS have shown that functional connectivity measured by both EEG and fMRI decreases when symptoms of MdDS improve. This study seeks to use asynchronous visual and auditory stimulation provided through a smart-phone app (WAVES) administered through virtual reality goggles to modulate the vertigo in MdDS with the hypothesis that these stimuli can desynchronize functional connectivity.

DETAILED DESCRIPTION:
The main device class used in this study will be an app that was designed by one of the investigators. The app is called "WAVES" and can be run on either an Android or iOS platform. The program presents a split screen of flashing lights with a different frequency on each half screen. The frequency of the lights can be changed according to either standard parameters or parameters set by EEG metrics. Audio stimulation will also be added in a second phase of the study. The audio stimulation consists of clicks given to each ear at different frequencies.

The study will have several stages. The participants will be told what stage of the project they will be participating in.

Stage 1: Open-label feasibility-this stage will include about 10-15 individuals who will be test participants for new protocols. This may include change in frequency of stimulation around a new baseline such as the individual theta frequency or the individual alpha frequency. All session parameters will be restricted, e.g. no more than 40-minutes of total stimulation per session.

Stage 2: Sham controlled single-blind randomized onsite. This stage will include participants who receive up to 40-minutes of visual stimulation given either through a protocol determined in Stage 1 as an effective paradigm or as random frequency stimulation. The participants will be blinded to study allocation. The principal investigator will not be blinded in order to have tighter oversight on safety.

Stage 3: Sham controlled double-blind randomized at home with cross over study. This stage will involve sending the participants home with a smartphone app and pre-fitted head mounted virtual reality frame. The participants will receive a kit that contains the accessories and smartphone. Allocation will be 1:1 real to sham stimulation. After a preset trial duration (generally 2-weeks) the participants who were give sham stimulation will be cross-overed to real stimulation. The individuals who underwent real stimulation will be cross-overed to sham stimulation for 2 weeks. Both will then be given the option of doing 2 weeks of open label stimulation and then tapered to off over 2 weeks. This will provide an assessment of stimulation efficacy of 2 weeks vs 4 weeks as well as the sham response rate. Each week of sessions entails 5-10 sessions per week.

The participants will be completing online study questionnaires through a personalized weblink on RedCap or SurveyMonkey.

EEG recordings will be made at baseline, conclusion, and in between sessions to monitor the correlation between symptoms and EEG features.

ELIGIBILITY:
Inclusion Criteria:

* 1. Persistent oscillating vertigo that occurs within 48-hours of disembarking from a moving vessel such as a boat, car, or plane, 2. Symptoms improve with exposure to passive motion, 3. No other cause for symptoms after evaluation by a neurologist or otolaryngologist.

Exclusion Criteria:

* 1. History of epilepsy. 2. Structural brain injury such as stroke, brain tumor, or confluent white matter lesions. 3. Unstable medical or psychiatric condition. 4. Pregnant or planning to become pregnant during the study duration. 5. Not able to comply with all study procedures.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2023-03-01 (Estimated); Primary Completion 2026-12 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
MdDS Balance Rating Scale (MBRS) | 5 years
  This is a 10 point self-reported scale that assesses the severity of rocking dizziness and its effect on balance function. The scale goes from 1 to 10 with 1 representing no feeling of motion and 10 representing motion severity so strong that standing is not possible.

SECONDARY OUTCOMES:
Visual Analogue Scale | 5 years
  100 point scale of global assessment of MdDS related symptoms. This scale goes from 0 to 100 with 0 representing no symptoms attributable to MdDS at all and 100 representing global symptom severity due to MdDS so severe that one is completely not functional. This scale takes into account the other symptoms of MdDS besides the feeling of motion. These other symptoms could be cognitive slowing, fatigue, visual motion intolerance, headache, and anxiety.
Hospital Anxiety Depression Scale | 5 years
  A 14 item inventory of depression and anxiety symptoms that has separate items that assess depression and anxiety. Each item has a maximum of 3 possible points with higher values representing higher symptom severity. There are 21 possible points for depression and 21 possible points for anxiety.
Dizziness Handicap Inventory | 5 years
  This is a standardized assessment of dizziness with items inquiring about physical, emotional, and functional elements. There are 25 questions that can each be scored up to 4 points with higher scores representing more severe symptoms.

OTHER OUTCOMES:
Electroencephalography (EEG) | 5 years
  EEG is a method to measure brain electrical activity. This activity has frequency components (theta, alpha, beta, etc.). Those frequency components can be used to measure functional connectivity between different brain regions by examining how much these components are in sync. The connectivity changes can be different across frequencies and brain regions. Functional connectivity measured by EEG as a function of symptom change and stimulation frequency will be an exploratory outcome of the study.

CONTACTS AND LOCATIONS:
Overall Officials: Yoon-Hee Cha, MD, Principal Investigator — University of Minnesota

IPD SHARING:
Plan to Share IPD: Yes
Study protocol and de-identified data may be shared with through an institutional data sharing agreement.
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: 5 years
Access Criteria: Well-established or working under the supervision of a well-established researcher in the neurosciences with adequate justification for accessing the data under an appropriate data sharing agreement.